CLINICAL TRIAL: NCT00868634
Title: Capecitabine and Bevacizumab ± Vinorelbine as 1st Line Treatment in HER-2 Negative Metastatic or Locally Advanced Inoperable Breast Cancer Patients
Brief Title: Capecitabine and Bevacizumab ± Vinorelbine in Metastatic Breast Cancer
Acronym: CARIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: iOMEDICO AG (Industry)
Collaborators: Arbeitsgemeinschaft fur Internistische Onkologie (Other); Arbeitskreis Klinische Studien (Other); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOM-080-2; 2008-003779-37 (EudraCT Number)
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Bevacizumab; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Capecitabine / Bevacizumab
  Interventions: Drug: capecitabine; Drug: bevacizumab
- B (Experimental): Capecitabine / Bevacizumab / Vinorelbine
  Interventions: Drug: capecitabine; Drug: bevacizumab; Drug: vinorelbine

INTERVENTIONS:
Drug: capecitabine — 1000 mg/m2 twice daily, oral, days 1-14. Cycles are repeated every three weeks.
  Other Names: Xeloda®
  Arms: A
Drug: bevacizumab — 15 mg/kg i.v., day 1 Cycles are repeated every three weeks.
  Other Names: Avastin®
  Arms: A
Drug: capecitabine — 1000 mg/m2 twice daily, oral, days 1-14. Cycles are repeated every three weeks.
  Other Names: Xeloda®
  Arms: B
Drug: bevacizumab — 15 mg/kg i.v., day 1. Cycles are repeated every three weeks.
  Other Names: Avastin®
  Arms: B
Drug: vinorelbine — 25 mg/m2 i.v., days 1+8. Cycles are repeated every three weeks.
  Other Names: Navirel®
  Arms: B

SUMMARY:
The aim of the trial is to detect the superiority of the triple combination of capecitabine, bevacizumab and vinorelbine versus the combination of capecitabine and bevacizumab in patients with metastatic breast cancer. 600 patients, 300 in each treatment group, are treated until progression of disease to determine PFS.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent.
* Able to comply with the protocol.
* ECOG Performance status 0 - 2.
* Life expectancy more than 12 weeks.
* Known ER / PR status.
* Confirmed HER2/neu-negative, adenocarcinoma of the breast with measurable or non-measurable locally recurrent or metastatic disease, who are candidates for chemotherapy.
* Previous (neo)adjuvant chemotherapy is allowed provided that the last dose of chemotherapy was applied more than 6 months prior to randomization.
* Previous adjuvant radiotherapy is allowed as part of the treatment of early breast cancer provided that no more than 30% of marrow-bearing bone was irradiated.
* No signs and symptoms of CHF.
* Adequate hepatic and renal function values.
* Adequate hematologic function values.

Key Exclusion Criteria:

* Pregnant or lactating females.
* Previous chemotherapy for metastatic or locally recurrent breast cancer.
* Previous radiotherapy for the treatment of metastatic disease (unless given for the relief of metastatic bone pain)
* Evidence of spinal cord compression or current evidence of central nervous system (CNS) metastases.
* Major surgical procedure, open biopsy or significant traumatic in-jury within 28 days prior to randomization, or anticipation of the need for major surgery during the course of the study treatment.
* History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding.
* Uncontrolled hypertension (systolic > 150 mmHg and/or diastolic > 100 mmHg). Clinically significant (i.e. active) cardiovascular disease, requiring medication during the study and might interfere with regularity of the study treatment, or not controlled by medication.
* Non-healing wound, active peptic ulcer or bone fracture.
* History of abdominal fistula, or any grade 4 nongastrointestinal fistula, gastrointestinal perforation or intrabdominal abscess within 6 months of randomization.
* Active infection requiring i.v. antibiotics at randomization.
* Clinically significant malabsorption syndrome or inability to take oral medication.
* Known hypersensitivity to any of the study drugs or excipients.
* Concurrent treatment with any drug interfering with study medication. Concurrent participation in another clinical trial. Prior participation is allowed when the last study medication was applied more than 4 weeks prior to randomization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2009-02; Primary Completion 2014-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | end of trial

SECONDARY OUTCOMES:
adverse events and serious adverse events | during the whole time of treatment
Overall Response Rate (ORR = CR +PR) | end of trial
Overall Survival (OS) | end of trial

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Hegewisch-Becker, MD, Principal Investigator — Onkologische Schwerpunktpraxis Eppendorf
Locations (1):
- Onkologische Schwerpunktpraxis Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No